CLINICAL TRIAL: NCT04120220
Title: Shake It Up: Lipidomics of Lipoproteins and Diet
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI will be retiring from the Center. Research will not continue with a new PI.
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GFHNRC511
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Overweight
Keywords: Normal weight
MeSH Terms: conditions — Overweight | interventions — Soybean Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy Cream (Experimental): Participants will receive a meal containing 30 g of fat prepared with heavy cream.
  Interventions: Other: Heavy Cream
- Soybean Oil (Experimental): Participants will receive a meal containing 30 g of fat prepared with soybean oil.
  Interventions: Other: Soybean Oil

INTERVENTIONS:
Other: Heavy Cream — Participants will receive a meal in the form of a fruit-containing shake containing 30 g of fat prepared with heavy cream.
  Arms: Heavy Cream
Other: Soybean Oil — Participants will receive a meal in the form of a fruit-containing shake containing 30 g of fat prepared with soybean oil.
  Arms: Soybean Oil

SUMMARY:
The purpose of this research is to understand how dietary fat is related to cardiovascular disease (CVD). This study tests the effect of different dietary fats on the level of fat in the blood and the particles that transport fat in the blood. The researchers want to know if these particles change after eating meals made with different fats.

DETAILED DESCRIPTION:
The overall objective of this work is to discover how the lipidomic composition of postprandial lipoproteins responds to dietary fats of differing fatty acid composition by comparing meals rich in saturated fatty acid (SFA) (from dairy cream) versus polyunsaturated fatty acids (PUFA) (from soybean oil). The information derived from these studies will provide mechanistic insight into postprandial lipid metabolism and will support efforts to identify optimal dietary oil intakes for people.

ELIGIBILITY:
Inclusion Criteria:

* Normal to overweight (BMI 18.0-29.9 kg/m^2
* Willing to comply with the demands of the experimental protocol

Exclusion Criteria:

* Inability to provide consent
* Have fasting blood glucose <60 mg/dL or >126 mg/dL
* Have fasting blood cholesterol >300 mg/dL
* Have fasting blood triglyceride <100 mg/dL or >300 mg/dL
* Have uncontrolled hypertension (blood pressure >140/90 mm Hg)
* Take prescription medications for blood sugar or lipid management or anti-inflammatory steroids (e.g. cortisone)
* Over the counter use of supplements (fish oil, flax, plant sterol or sterol esters) and unwilling to discontinue use for 6 weeks prior to study initiation
* Have a history of an eating disorder, unusual dietary pattern (extreme nutrient or food group restriction; erratic meals due to shift work, etc.)
* Have established cardiovascular, pulmonary, and/or a metabolic disease such as diabetes
* Have cancer
* Use tobacco products or nicotine in any form including snuff, pills, and patches, or e-cigarettes/vaping in the past 6 weeks
* Have alcohol, anabolic steroids, or other substance abuse issues
* Consume more than 3 alcoholic drinks/week
* Are lactose intolerant or have an allergy to dairy foods

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
Change in lipidomic composition of plasma post-prandial lipoproteins as assessed by incremental area under the curve (iAUC) | 0, 1, 2, 4, 6, 8 hours post meal intake

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Picklo, PhD, Principal Investigator — USDA Grand Forks Human Nutrition Research Center
Locations (1):
- USDA Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Grand Forks Human Nutrition Research Center Current Nutrition Studies — https://www.ars.usda.gov/plains-area/gfnd/gfhnrc/docs/nutrition-studies/nutrition-studies/

DOCUMENTS (1):
  • Informed Consent Form (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT04120220/ICF_000.pdf